CLINICAL TRIAL: NCT03442751
Title: A Phase III, Multi-center Study to Evaluate the Safety and Efficacy of Epithelium-on Corneal Collagen Cross-linking in Eyes With Progressive Keratoconus
Brief Title: Study to Evaluate the Safety and Efficacy of Epi-on Corneal Cross-linking in Eyes With Progressive Keratoconus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-KXL-308
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Progressive Keratoconus

STUDY DESIGN:
Intervention Model Description: Randomization was by eye (active or sham). However an individual participant could receive active/active, active/untreated, sham/sham, sham/untreated or active/sham
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Epithelium-on CXL Treatment Group (Experimental): Study eye receives Test Article A, Test Article B, and exposed to cross-linking dose of UVA light generated by the KXL medical device system
  Interventions: Drug: Test Article A; Drug: Test Article B; Device: KXL medical device system
- Sham Treatment/Control Group (Sham Comparator): Sham eye receives Placebo and and exposed to mock dose of UVA light generated by the KXL medical device system
  Interventions: Drug: Placebo; Device: KXL medical device system

INTERVENTIONS:
Drug: Test Article A — Riboflavin Ophthalmic Solution A
  Arms: Epithelium-on CXL Treatment Group
Drug: Test Article B — Riboflavin Ophthalmic Solution B
  Arms: Epithelium-on CXL Treatment Group
Drug: Placebo — Placebo Vehicle of Test Article
  Arms: Sham Treatment/Control Group
Device: KXL medical device system — Mock UVA light source
  Arms: Sham Treatment/Control Group
Device: KXL medical device system — Cross-linking UVA light source
  Arms: Epithelium-on CXL Treatment Group

SUMMARY:
To evaluate the safety and efficacy of epithelium-on corneal collagen cross-linking (CXL) in impeding the progression of, and/or reducing corneal curvature (Kmax) in eyes with progressive keratoconus. Epithelium-on CXL uses a formulation that allows the riboflavin to penetrate the cornea without the need to remove the epithelium, the outer most layer of the cornea.

DETAILED DESCRIPTION:
Up to 275 study eyes with progressive keratoconus will be enrolled. Study eyes will be randomized in a 2:1 ratio to receive CXL treatment or sham/control treatment.The primary efficacy endpoint is a difference of ≥ 1 diopter between treatment groups in the mean change in Kmax from baseline to Month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 12 and 55 years of age, male or female, of any race;
2. Provide written informed consent and sign a HIPAA form. Subjects who are under the age of 18 (or have not yet reached the age of majority per local regulations) will need to sign an assent form as well as having a parent or legal guardian sign an informed consent
3. Ability to read English or Spanish to complete the NEI-VFQ 25 questionnaire;
4. Willingness and ability to follow all instructions and comply with schedule for follow-up visits;
5. For females capable of becoming pregnant, agree to have urine pregnancy testing performed prior to randomization of each study eye; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the randomization visit, and continue to use the method for one month following the treatment. Acceptable forms for birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (e.g. hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
6. Having topographic and clinical evidence of keratoconus

Exclusion Criteria:

1. Contraindications, sensitivity or known allergy to the use of the test article(s) or their components;
2. If female, be pregnant, nursing or planning a pregnancy or have a positive urine pregnancy test prior to the randomization or treatment of either eye or during the course of the study;
3. Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications.
4. A history of delayed epithelial healing in the eye to be treated or a current condition that may interfere with or prolong epithelial healing;
5. A history of previous corneal cross-linking treatment in the eye to be treated;
6. Have used an investigational drug or device within 30 days of screening or be concurrently enrolled in another investigational drug or device trial within 30 days of the study.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 201 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Smith, Study Director — Glaukos Corporation
Locations (1):
- Ophthalmic Consultants of Boston, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at eye clinics and were required to meet inclusion/exclusion criteria prior to enrollment
Pre-assignment Details: 280 eyes of 201 subjects were randomized in a 2:1 treatment allocation. Of the 280 randomized eyes, 279 were treated: 189 eyes of 156 subjects received CXL treatment & 90 eyes of 83 subjects received Sham/Control, for a total of 239 treatments. Of the 201 unique subjects, 118 received CXL only (in 1 or both eyes), 45 received Sham/Control only (in 1 or both eyes), and 38 subjects received CXL in 1 eye and Sham/Control in the other eye.
Units Other Than Participants: eyes
Groups:
- Epithelium-on CXL Treatment Group: Study eye receives riboflavin ophthalmic solution A, riboflavin ophthalmic solution B and irradiated using KXL High Power System Riboflavin Ophthalmic Solution A Riboflavin Ophthalmic Solution B: KXL High Power System
- Sham Treatment/Control Group: Sham eye receives Placebo (the vehicle of Riboflavin Ophthalmic Solution) and Mock UVA light source
  Placebo KXL High Power System providing mock UVA light source
Period: Overall Study
Arm/Group | Epithelium-on CXL Treatment Group | Sham Treatment/Control Group
Started | 156; 189 eyes | 83; 90 eyes
Month 6 | 153; 186 eyes | 82; 89 eyes
Month 12 | 150; 183 eyes | 0; 0 eyes
Completed | 150; 183 eyes | 82; 89 eyes
Not Completed | 6; 6 eyes | 1; 1 eyes
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with progressive keratoconus in at least one eye (study eye). Subjects may contribute more than one eye if both eyes qualify. Eyes vs. subjects were randomized to the treatment arms.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Epithelium-on CXL Treatment Group | Sham Treatment/Control Group | Total
Number analyzed (Participants) | 156 | 83 | 201
Number analyzed (Eyes) | 189 | 90 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (9.75) | 29.5 (9.67) | 30.0 (9.9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 109 | 55 | 139
  Female | 47 | 28 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnicity: Hispanic or Latino | 28 | 68 | 36
  Ethnicity: Not Hispanic or Latino | 128 | 15 | 165
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Asian | 3 | 4 | 5
  Race: Black or African American | 27 | 18 | 36
  Race: Native Hawaiian or Other Pacific Islander | 3 | 1 | 3
  Race: White | 112 | 54 | 142
  Race: Other | 11 | 6 | 15
Mean Kmax (D) [Mean (Standard Deviation); unit: Diopters] — Kmax = maximal corneal curvature of the study eye(s)
  Diopters | 59.4 (9.1) | 59.3 (9.1) | 59.4 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Treatment Groups in the Change From Baseline to Month 6 in Kmax
Description: Mean difference of at least 1 diopter in Kmax change from baseline to Month 6 between treatment groups
Time Frame: 6 months
Population: Intent-to-treat analysis set which included all randomized study eyes that had at least one post-treatment follow-up efficacy assessment. Missing post-baseline Kmax data were imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Epithelium-on CXL Treatment Group | Sham Treatment/Control Group
Number analyzed (Participants) | 156 | 83
Number analyzed (eyes) | 189 | 90
Diopters | -0.3 [-0.6 to -0.0] | 0.6 [0.2 to 1.1]
Statistical Analysis 1: Comparison: Epithelium-on CXL Treatment Group vs Sham Treatment/Control Group; Repeated measures mixed analysis of covariance model; Test type: Superiority; p = 0.0004, ANCOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.5 to -0.4]

2. Secondary Outcome: Difference Between Treatment Groups in the Change From Baseline to Month 12 in Kmax
Description: Difference between the CXL and Sham/Control treatment groups in the change from baseline to Month 12 in Kmax
Time Frame: 12 months
Population: Intent-to-treat analysis set which included all randomized study eyes that had at least one post-treatment follow-up efficacy assessment. Missing post-baseline Kmax data were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Epithelium-on CXL Treatment Group | Sham Treatment/Control Group
Number analyzed (Participants) | 156 | 83
Number analyzed (eyes) | 189 | 90
Diopters | -0.4 [-0.7 to -0.2] | 0.7 [0.3 to 1.1]
Statistical Analysis 1: Comparison: Epithelium-on CXL Treatment Group vs Sham Treatment/Control Group; repeated measures mixed analysis of covariance model; Test type: Superiority — last observation carried forward was used to impute missing Month 12 data; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.1, 95% CI 2-sided [-1.6 to -0.6]

ADVERSE EVENTS:
Time Frame: 12 months for the Epithelium-on CXL Treatment Group and 6 months for the Sham Treatment/Control Group
Description: For the ocular adverse event arms, the affected and at risk population reflect the number of eyes.
  For the non-ocular adverse event arms, the affected and at risk population reflect the number of participants.
Groups:
- Ocular: Epithelium-on CXL Treatment Group: Study eye received riboflavin ophthalmic solution A, riboflavin ophthalmic solution B and irradiated using KXL High Power System
- Ocular: Sham Treatment/Control Group: Sham eye received Placebo (the vehicle of Riboflavin Ophthalmic Solution) and Mock UVA light source
- Non-ocular: Epithelium-on: Participant eye(s) treated only with this intervention (i.e., riboflavin ophthalmic solution A, riboflavin ophthalmic solution B and irradiated using KXL High Power System)
- Non-ocular: Sham Treatment/Control: Participant eye(s) treated only with this intervention (i.e., Placebo [the vehicle of riboflavin ophthalmic solution] and Mock UVA light source)
- Non-ocular: Epithelium-on and Sham Treatment: Participant had one eye treated with Epithelium-on CXL (i.e., riboflavin ophthalmic solution A, riboflavin ophthalmic solution B and irradiated using KXL High Power System) and one eye treated with Sham (i.e., Placebo [the vehicle of riboflavin ophthalmic solution] and Mock UVA light source)
Arm/Group | Ocular: Epithelium-on CXL Treatment Group | Ocular: Sham Treatment/Control Group | Non-ocular: Epithelium-on | Non-ocular: Sham Treatment/Control | Non-ocular: Epithelium-on and Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/90 | 0/118 | 0/45 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/189 | 0/90 | 2/118 | 0/45 | 1/38
Other Adverse Events (participants affected / at risk) | 170/189 | 63/90 | 1/118 | 0/45 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ocular: Epithelium-on CXL Treatment Group (N=189) | Ocular: Sham Treatment/Control Group (N=90) | Non-ocular: Epithelium-on (N=118) | Non-ocular: Sham Treatment/Control (N=45) | Non-ocular: Epithelium-on and Sham Treatment (N=38)
Urinary tract infection (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — posterior stromal haze post-operatively
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocular: Epithelium-on CXL Treatment Group (N=189) | Ocular: Sham Treatment/Control Group (N=90) | Non-ocular: Epithelium-on (N=118) | Non-ocular: Sham Treatment/Control (N=45) | Non-ocular: Epithelium-on and Sham Treatment (N=38)
Conjunctival hyperaemia (Eye disorders) | 115 (120) | 25 (27) | 0 (0) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 77 (97) | 11 (11) | 0 (0) | 0 (0) | 0 (0) — corneal haze
Photophobia (Eye disorders) | 73 (90) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 66 (84) | 27 (30) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 61 (70) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 59 (66) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 36 (37) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal epithelium defect (Eye disorders) | 28 (34) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal striae (Eye disorders) | 26 (27) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 22 (23) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 20 (21) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Anterior chamber flare (Eye disorders) | 20 (21) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 18 (20) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 18 (18) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 18 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal warpage (Eye disorders) | 13 (14) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 11 (12) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Corneal thinning (Eye disorders) | 11 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anterior chamber cell (Eye disorders) | 10 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vital dye staining cornea present (Investigations) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — corneal fluorescein staining
Eyelid oedema (Eye disorders) | 27 (27) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03442751/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03442751/SAP_001.pdf